CLINICAL TRIAL: NCT02578862
Title: Total Intravenous Versus Inhaled Anesthesia in Endoscopic Sinus Surgery for High-Grade Paranasal Disease
Brief Title: Total Intravenous Anesthesia in Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Edward Mccoul, MD, Active Medical Staff, Ochsner Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015.131.A
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-11

CONDITIONS: Advanced Chronic Rhinosinusitis
MeSH Terms: interventions — Propofol; Sevoflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total Intravenous (Experimental): Intravenous propofol for maintenance of anesthesia
  Interventions: Drug: Propofol
- Inhaled Anesthetic (Active Comparator): Inhaled volatile anesthetic for maintenance of anesthesia
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol
  Arms: Total Intravenous
Drug: Sevoflurane
  Other Names: Isoflurane
  Arms: Inhaled Anesthetic

SUMMARY:
Utilization of total intravenous anesthesia (TIVA) has been proposed as a method to improve visualization during endoscopic sinus surgery (ESS), largely due to its physiologic decrease in cardiac output without the peripheral smooth muscle relaxation and resultant vasodilation associated with inhaled anesthetics. This may be especially important in cases of advanced inflammatory sinus disease, when visualization may be most compromised. The goal of this study is to improve clinical practice paradigms by evaluating the use of TIVA versus inhaled anesthetic for maintenance of anesthesia in ESS for advanced paranasal sinus disease.

DETAILED DESCRIPTION:
Specific Aims:

1. Determine the effect of total intravenous versus inhaled anesthesia on intraoperative visual field in endoscopic sinus surgery for advanced paranasal sinus disease
2. Evaluate clinical outcomes associated with choice of total intravenous versus inhaled anesthesia in endoscopic sinus surgery

General Design:

Double blind, randomized controlled trial of total intravenous versus inhaled anesthetic for maintenance of anesthesia during endoscopic sinus surgery.

Subject Recruitment and Screening:

Patients will be screened for study inclusion by the principal investigator (EDM) during their preoperative visit in the Department of Otolaryngology. Those meeting inclusion criteria will be introduced to the study at this time. A full description of the research purpose, personnel, procedures, risks and benefits will be presented, and a copy of the study consent documentation will be provided for home review.

Method for Assigning Subjects to Treatment Groups:

On the day of surgery, eligible participants will be admitted to the Day of Surgery Department, where a member of the Anesthesia team will review study information and confirm informed consent. A randomly assigned, sealed envelope will then be opened to assign participants to either the TIVA, or inhaled anesthetic cohort. At no time will the patient or surgeon be made aware of the patient's cohort.

Blinding of Study Drug:

At no time will the patient or surgeon be made aware of the patient's cohort. During the procedure the surgeon is blinded to the type of anesthesia by placement of a high drape at the head of the operative table. Study reviewers will be blinded to treatment arm without cohort assignment at time of review for determination of visual field score.

Study Procedures:

Participants make no clinic/hospital visits for purposes of study completion as all patient interaction limited to visits and surveys completed as part of routine clinical care. Clinic visits will include a baseline preoperative visit, and visits at 1 week, 4 weeks, and 10 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endoscopic sinus surgery
* Advanced inflammatory sinus disease, defined as allergic fungal sinusitis, chronic rhinosinusitis with nasal polyposis, chronic rhinosinusitis with eosinophilia, or rhinosinusitis with pan-sinus opacification (Lund-Mackay score >12).

Exclusion Criteria:

* Noninflammatory sinonasal disease
* Disease extending through the skull base or orbital wall
* American Society of Anesthesiologists Preoperative Health Status >II
* Known non-pharmacologic coagulopathy (platelet < 50000/mL, international normalized ratio > 1.2)
* Preoperative anticoagulants within 7 days of surgery
* Allergy to one of the study medications
* Age under 18 years
* Non-English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward D McCoul, MD,MPH, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Brunner JP, Levy JM, Ada ML, Tipirneni KE, Barham HP, Oakley GM, Cox DR, Nossaman BD, McCoul ED. Total intravenous anesthesia improves intraoperative visualization during surgery for high-grade chronic rhinosinusitis: a double-blind randomized controlled trial. Int Forum Allergy Rhinol. 2018 Oct;8(10):1114-1122. doi: 10.1002/alr.22173. Epub 2018 Jul 6. PMID 29979837

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Intravenous: Intravenous propofol for maintenance of anesthesia
  Propofol
- Inhaled Anesthetic: Inhaled volatile anesthetic for maintenance of anesthesia
  Sevoflurane
Period: Overall Study
Arm/Group | Total Intravenous | Inhaled Anesthetic
Started | 37 | 35
Completed | 37 | 33
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Unplanned unilateral procedure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Intravenous | Inhaled Anesthetic | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 45 [20 to 77] | 55 [25 to 81] | 51.5 [35.3 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 21 | 24 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 37 | 35 | 72
Body Mass Index (BMI) [Mean (Inter-Quartile Range); unit: kg/m^2] | 31 [21 to 56] | 28 [19 to 53] | 29.1 [25.9 to 34.6]
American Society of Anesthesiologists (ASA) Physical Status [Count of Participants; unit: Participants] — ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    I | 2 | 3 | 5
    II | 28 | 25 | 53
    III | 7 | 7 | 14
Disease Factors [Number; unit: participants]
  Polyposis | 31 | 33 | 64
  Tissue Eosinophilia | 28 | 30 | 58
  Allergic Fungal Rhinosinusitis (AFRS) | 5 | 3 | 8
  Aspirin Exacerbated Respiratory Disease (AERD) | 3 | 3 | 6
Patient Assessments [Median (Inter-Quartile Range); unit: units on a scale] — Lund Mackay Score- measures sinus opacification, Min 0 Max 24. Higher score indicates more opacification.
  SNOT-22 Score (Sinonasal Outcome Test-22)- measures sinus symptoms. Min 0 Max 110. Higher score indicates worse symptoms.
  units on a scale
    Lund-Mackay Score | 14 [13 to 16] | 15 [13 to 20] | 14 [13 to 18]
    SNOT-22 Score (Baseline) | 48 [37 to 59] | 45.5 [27 to 58] | 47 [34 to 58]
Co-morbidities [Number; unit: participants]
  Systemic Hypertension | 16 | 13 | 29
  Diabetes Mellitus | 2 | 3 | 5
  Reactive Airway Disease | 16 | 16 | 32
  Coronary Artery Disease | 1 | 1 | 2
  Renal Disease | 0 | 2 | 2
  Non-sinus Dysrhythmias | 0 | 1 | 1
  Congestive Heart Failure | 1 | 0 | 1
  Tobacco Use | 8 | 13 | 21
  Chronic Obstructive Pulmonary Disease (COPD) | 3 | 4 | 7
  Peripheral Vascular Disease | 3 | 1 | 4
  Liver Disease | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Visual Field Assessment
Description: Wormald Visualization Scale (validated)
  Grade Assessment (0-10) -Higher scores indicate worsening visualization
  0 No bleeding
  1. 1-2 points of ooze
  2. 3-4 points of ooze
  3. 5-6 points of ooze
  4. 7-8 points of ooze
  5. 9-10 points of ooze (sphenoid fills in 60 seconds)*
  6. 10 points of ooze, obscuring surface (sphenoid fills in 50 seconds)*
  7. Mild bleeding/oozing from entire surgical surface with slow accumulation of blood in the post nasal space (sphenoid fills by 40 seconds)
  8. Moderate bleeding from entire surgical surface with moderate accumulation of blood in the post nasal space at (sphenoid fills by 30 seconds)
  9. Moderately severe bleeding with rapid accumulation of blood in the post nasal space (sphenoid fills by 20 seconds)
  10. Severe bleeding with nasal cavity filling rapidly(sphenoid fills in10 seconds)
Time Frame: Performed intraoperatively at the end of surgical case
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Total Intravenous | Inhaled Anesthetic
Number analyzed (Participants) | 37 | 35
units on a scale
  Right Frontal | 3.3 [2.0 to 4.3] | 4.3 [2.8 to 5.6]
  Right Ethmoid | 3.3 [2.1 to 4.3] | 4.2 [3.3 to 5.9]
  Right Sphenoethmoidal Recess | 3.3 [2.7 to 4.3] | 4.8 [3.7 to 6.3]
  Right Choana | 2.7 [2.3 to 3.3] | 3.3 [2.2 to 5.0]
  Left Frontal | 3.3 [2.7 to 4.8] | 4.0 [3.3 to 5.3]
  Left Ethmoid | 3.3 [2.7 to 4.3] | 4.3 [3.3 to 6.3]
  Left Sphenoethmoidal Recess | 3.3 [2.3 to 4.3] | 4.3 [3.0 to 6.7]
  Left Choana | 3.0 [2.3 to 3.7] | 3.7 [2.7 to 5.0]

2. Secondary Outcome: Sinus-related Quality of Life
Description: Sinonasal Outcomes Test (SNOT-22) (validated)- measures sinus symptoms. Minimum 0 Maximum 110. Higher scores indicate worse sinus symptoms.
Time Frame: 3 months and 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Total Intravenous | Inhaled Anesthetic
Number analyzed (Participants) | 37 | 35
units on a scale
  3 months | 20.1 [12.6 to 27.6] | 14.2 [6.4 to 22.0]
  6 months | 21.5 [10.0 to 33.0] | 15.2 [5.9 to 24.6]

3. Secondary Outcome: Intraoperative Blood Loss
Description: Amount of blood loss (milliliters) during surgery
Time Frame: At time of surgery
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Total Intravenous | Inhaled Anesthetic
Number analyzed (Participants) | 37 | 35
mL | 200 [100 to 450] | 300 [200 to 500]

4. Secondary Outcome: Surgical Time
Description: Total time spent in surgery (hours)
Time Frame: At time of surgery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Total Intravenous | Inhaled Anesthetic
Number analyzed (Participants) | 37 | 35
hours | 3.4 [2.9 to 3.9] | 3.4 [2.8 to 4.0]

5. Secondary Outcome: Post-anesthesia Care Unit Recovery Time
Description: Hours spent in post-anesthesia care unit post-operatively
Time Frame: Immediately following surgery (postoperative day zero)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Total Intravenous | Inhaled Anesthetic
Number analyzed (Participants) | 37 | 35
hours | 1.3 [1.0 to 1.6] | 1.7 [1.2 to 2.5]

6. Secondary Outcome: Number of Patients Treated With Post-operative Anti-emetics
Description: patients receiving medication for post-operative nausea and/or vomiting
Time Frame: 24 hours following surgery completion
Measure: Count of Participants; unit: Participants
Arm/Group | Total Intravenous | Inhaled Anesthetic
Number analyzed (Participants) | 37 | 35
Participants | 27 | 20

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Total Intravenous | Inhaled Anesthetic
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 0/37 | 0/35

LIMITATIONS AND CAVEATS:
By limiting study inclusion to Chronic Rhinosinusitis patients with bilateral nasal polyps and preoperative Lund-Mackay scores >12, we limit the generalizability of study findings. Single-site design limits external validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT02578862/Prot_SAP_000.pdf